CLINICAL TRIAL: NCT03310918
Title: Randomized Trial of a Collaborative Palliative and Leukemia Care Model for Patients With AML and MDS Receiving Non-Intensive Therapy
Brief Title: A Collaborative Palliative and Leukemia Care Model for Patients With AML and MDS Receiving Non-Intensive Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-327; ECOR grant 230593 (Other Grant/Funding Number: ECOR)
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS; Palliative care
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative palliative and oncology care (Experimental): * 1st palliative care visit within 30 days of randomization in the outpatient or hospital
  * In outpatient setting: once monthly palliative care visits (or video/ or phone)
  * During hospital admissions: At least twice weekly palliative care visits
  Interventions: Other: Palliative Care; Other: Standard Leukemia care
- Standard oncology care (Active Comparator): * Palliative care consults only upon request
  * Standard oncology care
  Interventions: Other: Standard Leukemia care

INTERVENTIONS:
Other: Palliative Care — Specialized medical care for people with serious illness. This type of care is focused on providing relief from the symptoms and stress of a serious illness. The goal is to improve quality of life for both the patient and the family
  Arms: Collaborative palliative and oncology care
Other: Standard Leukemia care — Standard care per the hospital guideline

SUMMARY:
This research study is evaluating the impact a collaborative palliative care and oncology team will have on end-of-life outcomes, quality of end-of-life care, and the quality of life, symptoms, and mood of patients with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) receiving non-intensive therapy

DETAILED DESCRIPTION:
Frequently people undergoing treatment for AML or MDS experience physical and emotional symptoms during the course of their illness. These can be very distressing to both patients and their caregivers. Patients with AML or MDS receiving non-intensive therapy also often experience a rapid decline in their health status and have a limited prognosis. Despite their limited life-expectancy, they rarely engage in discussion with their clinicians regarding their goals and preferences for care at the end of life. The study doctors want to know if the early introduction of a team of clinicians that specialize in the lessening (palliation) of many of these distressing symptoms and have expertise in enhancing communication about prognosis and illness trajectory may improve the overall care of patients with acute leukemia.

This team of clinicians is called the palliative care team and they focus on ways to improve the participant's pain and other symptom management (nausea, fatigue, shortness of breath, anxiety, etc.) and to assist the participant and the participant's caregivers in coping with the emotional and social issues associated with their diagnosis. The team consists of physicians and advance practice nurses who have been specially trained in the care of patients facing serious illness.

The main purpose of this study is to compare two types of care - standard oncology care and standard oncology care with collaborative involvement of palliative care clinicians to see which is better for improving the experience of patients with AML and MDS undergoing treatment.

The purpose of this research study is to find out whether introducing patients undergoing treatment for AML or MDS to the palliative care team can improve their end-of-life communication, understanding of their prognosis, and their physical and psychological symptoms during the course of their illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML receiving non-intensive therapy including hypomethylating agents, single-agent chemotherapy, targeted therapy agents, or single or combination non-intensive agents offered on a clinical trial, including the following populations:

  * Newly diagnosed AML
  * Relapsed AML
  * Primary refractory AML
* The ability to provide informed consent
* The ability to comprehend English or complete questionnaires with minimal assistance of an interpreter

Exclusion Criteria:

* Patients not receiving care at MGH
* Patients receiving intensive chemotherapy (requiring 4-6 week hospitalization)
* Patients receiving supportive care alone
* Major psychiatric illness or co-morbid conditions prohibiting compliance with study procedures
* Patients already receiving palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from documentation of end-of-life care preferences to death | up to 2 years
  comparison of time from documentation of end-of-life care preferences to death in the electronic health records

SECONDARY OUTCOMES:
Rates of documentation of end-of-life care preferences at least one week prior to death. | up to 2 years
  Comparison of the rate of documentation of end-of-life care preferences at least one week prior to death in the electronic health record
Patient-report of discussing end-of-life care preferences based on an item from the perception of treatment and prognosis questionnaire | up to 2 years
  comparison of patient-report of discussion end-of-life care preferences between the study arms
Compare Rate of hospitalization between the study arms | up to 30 days
  Compare rates of hospitalizations within 30 days of death between the study arms
Rate of hospice utilization and length-of-stay in hospice | up to 2 years
  Compare rates of hospice utilization and length-of-stay in hospice at the end of life between the study arms
compare quality of life | up to six months
  Compare quality of life (FACT-Leuk) at week-12 and longitudinally between the study arms. Score range 0-176 (higher scores indicating better quality of life)
compare symptom burden | up to six months
  Compare symptom burden (ESAS) at week-12 and longitudinally between the study arms. the ESAS score range 0-100 with higher scores indicating worse symptom burden.
compare mood | up to six months
  Compare change in mood (HADS) at week-12, and longitudinally between the study arms. HADS measures depression and anxiety symptoms (subscale range 0-21) higher scores indicating worse mood symptoms

OTHER OUTCOMES:
Rate of chemotherapy administration | up to 30 days prior to death
  compare rate of chemotherapy administration within 30 days of death between the two study arms
Rates of death in the hospital | up to 2 years
  compare rates of death in the hospital between the two study arms
caregiver-reported discussion of end-of-life care preferences as measured by the perception of treatment and prognosis questionnaire | one month
  compare caregiver-reported discussion of end-of-life care preferences between the study arms at one month
Compare quality of end-of-life care between the two study arms | up to 2 years
  compare quality of end-of-life care (FAMCARE) as reported by caregivers between the two study arms. FAMCARE score range 0-100, higher scores indicate better quality of end-of-life care

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen-Battaglia M, Sohn MB, Consagra W, Wang Y, Zhang Z, LoCastro M, Davis J, Buettner K, Mortaz S, El-Jawahri AR, Loh KP. Trajectories of physical well-being among adults with acute myeloid leukemia. Blood Adv. 2024 Jun 11;8(11):2612-2621. doi: 10.1182/bloodadvances.2023011804. PMID 38429079